CLINICAL TRIAL: NCT01129557
Title: Aldosterone Breakthrough During Diovan (Valsartan), Tekturna (Aliskiren), and Combination (Valsartan+Aliskiren) Anti-hypertensive Therapy in Patients With Proteinuric Kidney Disease
Brief Title: Aldosterone Breakthrough During Diovan, Tekturna, and Combination Therapy in Patients With Proteinuric Kidney Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Pietro Canetta, MD, Instructor in Clinical Medicine, Nephrology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAE0863; #IIRP-906 (Other: Novartis)
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-04

CONDITIONS: Proteinuric Kidney Disease; Diabetic Nephropathy; Hypertensive Nephrosclerosis; IgA Nephropathy; Focal Segmental Glomerulosclerosis; Glomerulopathy (Obesity-associated); Glomerulonephritis, Membranous
MeSH Terms: conditions — Diabetic Nephropathies; Glomerulonephritis, IGA; Glomerulosclerosis, Focal Segmental; Glomerulonephritis, Membranous | interventions — aliskiren; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tekturna (Active Comparator): Tekturna (Aliskiren), a direct renin inhibitor (DRI) 300 mg by mouth once daily for 9 months
  Interventions: Drug: Aliskiren
- Diovan (Active Comparator): Diovan (Valsartan), an angiotensin receptor blocker (ARB) 320 mg by mouth once daily for 9 months
  Interventions: Drug: Valsartan
- Tekturna & Diovan (Active Comparator): Tekturna (Aliskiren), a direct renin inhibitor (DRI) 150 mg by mouth once daily & Diovan (Valsartan), an angiotensin receptor (ARB) 160 mg by mouth once daily for 9 months
  Interventions: Drug: Aliskiren; Drug: Valsartan

INTERVENTIONS:
Drug: Aliskiren
  Other Names: Tekturna
  Arms: Tekturna; Tekturna & Diovan
Drug: Valsartan
  Other Names: Diovan
  Arms: Diovan; Tekturna & Diovan

SUMMARY:
Primary Hypothesis: Aldosterone breakthrough will occur at a far lower frequency during renin inhibition (0-10% over 9 months), alone or in combination with an ARB, compared to conventional ARB therapy (35-45% over 9 months). The investigators hypothesize that aldosterone breakthrough occurs due to accumulation of active precursor substances, most notably angiotensin II, produced in response to conventional RAAS blockade with ACEinhibitors and ARBs. The investigators believe that direct renin inhibition (DRI) should minimize this accumulation and therefore significantly lower or possibly eliminate the breakthrough effect.

Interruption of the renin-angiotensin-aldosterone system (RAAS) with angiotensin-converting enzyme inhibitors (ACE-Is) and angiotensin receptor blockers (ARBs), alone and in combination, has become a leading therapy to slow the progression of chronic heart and kidney disease. Both types of drugs inhibit the formation of aldosterone, a hormone, which has been shown to have harmful effects on patients with chronic heart and kidney disorders. This treatment is effective but not perfect since, even after an initial improvement, many patients become worse over the long term. This may be due to an unexpected increase in aldosterone, a phenomenon called "aldosterone breakthrough."

The purpose of this study is to find out whether the use of a direct renin inhibitor (DRI) alone, or in combination with an angiotensin receptor blocker (ARB), will lessen the occurrence of aldosterone breakthrough since direct renin inhibitors inhibit the formation of aldosterone at a very early step. This study will compare the effectiveness of adding Diovan (valsartan) or Tekturna (aliskiren) or a combination of Diovan and Tekturna to the usual antihypertensive treatment. The investigators will follow blood pressure, aldosterone levels, and urinary protein levels over 9 months to evaluate which of these therapies is most effective for treating hypertension in patients with proteinuric kidney disease.

DETAILED DESCRIPTION:
This is a randomized, open-label, three-arm study comparing Diovan (valsartan, an ARB), Tekturna (aliskiren, a DRI), and the combination of valsartan + aliskiren (i.e. ARB + DRI). One hundred twenty subjects (40 per arm) will be treated with Tekturna, Diovan, or a combination of both drugs for 9 months on top of their usual antihypertensive treatment. Changes in urinary aldosterone excretion will be monitored during therapy to measure the incidence of aldosterone breakthrough, defined as any sustained positive change from baseline urinary aldosterone excretion by the completion of the 9-month study period. This frequency measure will be compared during ARB, DRI, and ARB + DRI therapy. Changes in urinary protein excretion will also be monitored alongside the urinary aldosterone levels to determine whether aldosterone breakthrough is associated with refractory proteinuria. This is an innovative study that will be the first to (1) examine aldosterone breakthrough during DRI therapy, and (2) explore whether addition of a DRI to an ARB protects against aldosterone breakthrough. In addition, this will be the first study to examine whether DRI therapy (alone or in combination with ARB) is effective therapy for hypertension in patients with non-diabetic proteinuric kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Proteinuria > 300 mg/day
* Normal to mildly reduced kidney function (eGFR > 45 ml/min/1.73m2)
* Systolic blood pressure >130 mm Hg
* Diastolic blood pressure >70 mm Hg
* Diagnoses of diabetic nephropathy, hypertensive nephrosclerosis, IgA nephropathy, focal segmental glomerulosclerosis, membranoproliferative glomerulonephritis, membranous nephropathy, fibrillary glomerulonephritis, or obesity-associated glomerulopathy

Exclusion Criteria:

* Concomitant use of cyclosporine (which can interact with aliskiren)
* Inability to undergo 6 week washout period if already on RAAS-blocking drug(s) (includes renin inhibitor, ACE-inhibitor, ARB, and mineralocorticoid receptor blocker)
* eGFR < 45 ml/min/1.73m2
* Urine protein excretion < 300 mg/day
* Serum K > 5.0 mEq/l
* Systolic blood pressure > 170 mm Hg or < 130 mm Hg after washout period
* Diastolic blood pressure > 110 mm Hg or < 70 mm Hg after washout period
* Congestive heart failure NYHA class III and IV
* History of any cardiovascular events (stroke, TIA, MI, unstable angina, CABG, PCI, CHF hospitalization) in 3 months prior to study visit 1
* 2nd or 3rd degree heart block without a pacemaker or other uncontrolled arrhythmia
* Clinically significant valvular disease
* Known renal artery stenosis
* Any surgical or medical condition that might significantly alter the pharmacokinetics of the study drugs (n.b. bariatric surgery > 6 months prior to visit 1 is not an exclusion)
* History or evidence of drug or alcohol abuse within the last 12 months
* Any concurrent life threatening condition with a life expectancy less than 2 years
* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless postmenopausal for at least 1 year, surgically sterile, or using effective methods of contraception as defined by local health authorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Canetta, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Bomback AS, Rekhtman Y, Klemmer PJ, Canetta PA, Radhakrishnan J, Appel GB. Aldosterone breakthrough during aliskiren, valsartan, and combination (aliskiren + valsartan) therapy. J Am Soc Hypertens. 2012 Sep-Oct;6(5):338-45. doi: 10.1016/j.jash.2012.07.003. PMID 22995802

RESULTS

PARTICIPANT FLOW:
Groups:
- Tekturna + Diovan: Tekturna (Aliskiren), a direct renin inhibitor (DRI) 150 mg by mouth once daily for 9 months & Diovan (Valsartan), an angiotensin receptor blocker (ARB) 160 mg by mouth once daily for 9 months
Period: Overall Study
Arm/Group | Diovan | Tekturna | Tekturna + Diovan
Started | 15 | 17 | 14
Completed | 11 | 12 | 10
Not Completed | 4 | 5 | 4
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Novartis terminated study early | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Tekturna+Diovan: Tekturna (Aliskiren), a direct renin inhibitor (DRI) 150 mg by mouth once daily for 9 months & Diovan (Valsartan), an angiotensin receptor blocker (ARB) 160 mg by mouth once daily for 9 months
- Total: Total of all reporting groups
Arm/Group | Diovan | Tekturna | Tekturna+Diovan | Total
Number analyzed (Participants) | 15 | 17 | 14 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 12 | 44
  >=65 years | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 14
  Male | 11 | 11 | 10 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 8 | 8 | 9 | 25
  More than one race | 4 | 4 | 2 | 10
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Aldosterone Breakthrough in Subjects Who Completed the 9-month Study Protocol.
Description: The primary outcome of this study is the 9-month cumulative incidence of aldosterone breakthrough, defined as a sustained increase in 24-hour urine aldosterone above baseline, in each treatment arm.
Time Frame: 9 months
Measure: Number; unit: participants
Groups:
- Diovan: valsartan [angiotensin receptor blocker (ARB)] : Diovan 320 mg PO once daily for 9 months
- Tekturna: aliskiren [direct renin inhibitor (DRI)] : Tekturna 300 mg PO once daily for 9 months
- Tekturna + Diovan: aliskiren + valsartan (DRI + ARB) : Tekturna 150 mg PO once daily + Diovan 160 mg PO once daily for 9 months
Arm/Group | Diovan | Tekturna | Tekturna + Diovan
Number analyzed (Participants) | 11 | 12 | 10
participants | 3 | 3 | 3

2. Secondary Outcome: Serum Aldosterone Over Time During 9-month Treatment Course in Subjects With and Without Aldosterone Breakthrough.
Description: Mean serum aldosterone at baseline, 3-, 6-, and 9-months.
Time Frame: Baseline, 3-, 6-, and 9-months
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | 3 Months: Subjects Without Aldosterone Breakthrough | 6 Months: Subjects Without Aldosterone Breakthrough | 9 Months: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | 3 Months: Subjects With Aldosterone Breakthrough | 6 Months: Subjects With Aldosterone Breakthrough | 9 Months: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 9 | 9 | 9 | 9
ng/dL | 9.1 (5.2) | 4.8 (3.1) | 4.9 (3.6) | 4.9 (3.8) | 7.3 (4.5) | 8.5 (4.3) | 11.7 (5.6) | 11.7 (7.5)

3. Secondary Outcome: Urine Aldosterone Over Time During 9-month Treatment Course in Subjects With and Without Aldosterone Breakthrough.
Description: Mean urine aldosterone at baseline, 3-, 6-, and 9-months.
Time Frame: Baseline, 3-, 6-, and 9-months
Measure: Mean (Standard Deviation); unit: ug/day
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | 3 Months: Subjects Without Aldosterone Breakthrough | 6 Months: Subjects Without Aldosterone Breakthrough | 9 Months: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | 3 Months: Subjects With Aldosterone Breakthrough | 6 Months: Subjects With Aldosterone Breakthrough | 9 Months: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 9 | 9 | 9 | 9
ug/day | 10.9 (9.4) | 4.4 (3.3) | 5.5 (4.3) | 4.3 (2.3) | 7.4 (4.5) | 11.0 (6.2) | 14.4 (8.2) | 12.8 (5.2)

4. Secondary Outcome: Serum Potassium Over Time During 9-month Treatment Course in Subjects With and Without Aldosterone Breakthrough.
Description: Mean serum potassium at baseline, 3-, 6-, and 9-months. (given as reference to interpret contemporaneous plasma & urine aldosterone measurements.)
Time Frame: Baseline, 3-, 6-, and 9-months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | 3 Months: Subjects Without Aldosterone Breakthrough | 6 Months: Subjects Without Aldosterone Breakthrough | 9 Months: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | 3 Months: Subjects With Aldosterone Breakthrough | 6 Months: Subjects With Aldosterone Breakthrough | 9 Months: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 9 | 9 | 9 | 9
mmol/L | 4.2 (0.5) | 4.4 (0.5) | 4.4 (0.4) | 4.4 (0.4) | 4.3 (0.2) | 4.2 (0.2) | 4.3 (0.2) | 4.4 (0.4)

5. Secondary Outcome: Mean 24-hour Urine Sodium Over Time During 9-month Treatment Course in Subjects With and Without Aldosterone Breakthrough.
Description: Mean 24-hour urine sodium (mmol/day) at baseline, 3-, 6-, and 9-months. (given as reference to interpret contemporaneous plasma & urine aldosterone measurements.)
Time Frame: Baseline, 3-, 6-, and 9-months
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | 3 Months: Subjects Without Aldosterone Breakthrough | 6 Months: Subjects Without Aldosterone Breakthrough | 9 Months: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | 3 Months: Subjects With Aldosterone Breakthrough | 6 Months: Subjects With Aldosterone Breakthrough | 9 Months: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 9 | 9 | 9 | 9
mmol/day | 158 (67) | 180 (81) | 188 (66) | 169 (70) | 258 (98) | 220 (65) | 250 (102) | 200 (54)

6. Secondary Outcome: Pre- and Post-treatment Blood Pressure in Subjects With and Without Aldosterone Breakthrough.
Description: Compares baseline and final (9 month) blood pressure for subjects with and without aldosterone breakthrough
Time Frame: Baseline and Final (9 month)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | Final: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | Final: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 9 | 9
mm Hg
  Office systolic Blood Pressure | 134.0 (10.9) | 122.0 (12.0) | 136.3 (9.8) | 127.9 (10.8)
  Office diastolic Blood Pressure | 83.7 (8.9) | 74.0 (9.3) | 87.7 (6.6) | 81.6 (10.2)

7. Secondary Outcome: Pre- and Post-treatment Serum Creatinine in Subjects With and Without Aldosterone Breakthrough.
Description: Compares baseline and final (9 month) serum creatinine for subjects with and without aldosterone breakthrough
Time Frame: Baseline and Final (9 month)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | Final: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | Final: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 9 | 9
mg/dL | 1.2 (0.3) | 1.3 (0.4) | 1.2 (0.5) | 1.4 (1.1)

8. Secondary Outcome: Pre- and Post-treatment Serum Potassium in Subjects With and Without Aldosterone Breakthrough.
Description: Compares baseline and final (9 month) serum potassium for subjects with and without aldosterone breakthrough
Time Frame: Baseline and Final (9 month)
Measure: Mean (Standard Deviation); unit: (mmol/L)
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | Final: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | Final: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 9 | 9
(mmol/L) | 4.2 (0.5) | 4.4 (0.4) | 4.3 (0.2) | 4.4 (0.4)

9. Secondary Outcome: Pre- and Post-treatment 24-hour Urine Protein in Subjects With and Without Aldosterone Breakthrough.
Description: Compares baseline and final (9 month) 24-hour urine protein for subjects with and without aldosterone breakthrough
Time Frame: Baseline and Final (9 month)
Measure: Mean (Standard Deviation); unit: (mg/day)
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | Final: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | Final: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 9 | 9
(mg/day) | 2827 (2736) | 1911 (2958) | 3844 (3502) | 2681 (2967)

10. Secondary Outcome: Pre- and Post-treatment 24-hour Urine Sodium in Subjects With and Without Aldosterone Breakthrough.
Description: Compares baseline and final (9 month) 24-hour urine sodium for subjects with and without aldosterone breakthrough
Time Frame: Baseline and Final (9 month)
Measure: Mean (Standard Deviation); unit: (mmol/day)
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | Final: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | Final: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 9 | 9
(mmol/day) | 158 (67) | 169 (70) | 258 (98) | 200 (54)

11. Secondary Outcome: Pre- and Post-treatment 24-urine Aldosterone in Subjects With and Without Aldosterone Breakthrough.
Description: Compares baseline and final (9 month) 24-hour urine aldosterone for subjects with and without aldosterone breakthrough
Time Frame: Baseline and Final (9 month)
Measure: Mean (Standard Deviation); unit: (ug/day)
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | Final: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | Final: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 9 | 9
(ug/day) | 10.9 (9.4) | 4.3 (2.3) | 7.4 (4.5) | 12.8 (5.2)

12. Secondary Outcome: Pre- and Post-treatment Serum Aldosterone in Subjects With and Without Aldosterone Breakthrough.
Description: Compares baseline and final (9 month) serum aldosterone for subjects with and without aldosterone breakthrough
Time Frame: Baseline and Final (9 month)
Measure: Mean (Standard Deviation); unit: (ng/dL)
Arm/Group | Baseline: Subjects Without Aldosterone Breakthrough | Final: Subjects Without Aldosterone Breakthrough | Baseline: Subjects With Aldosterone Breakthrough | Final: Subjects With Aldosterone Breakthrough
Number analyzed (Participants) | 24 | 24 | 9 | 9
(ng/dL) | 9.1 (5.2) | 4.9 (3.8) | 7.3 (4.6) | 11.7 (7.5)

ADVERSE EVENTS:
Arm/Group | Tekturna | Diovan | Tekturna + Diovan
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 2/17 | 1/15 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tekturna (N=17) | Diovan (N=15) | Tekturna + Diovan (N=14)
>25% increase in creatinine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (General disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No